CLINICAL TRIAL: NCT03656484
Title: Innovative Technology for Assessing the Periodontal Disease and New Periodontitis Treatment Based on Hyaluronic Acid and Melatonin
Brief Title: New Periodontitis Treatment Based on Hyaluronic Acid and Melatonin
Acronym: HAMELDENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concordia Dent Srl (Other)
Collaborators: Carol Davila University of Medicine and Pharmacy (Other); Romanian National Authority for Scientific Research and Innovation (UEFISCIDI) (Unknown); University Politechnica of Bucharest (Unknown); TURKEY MEDISEN Ltd (Unknown)
Responsible Party: Principal Investigator, Corina Marilena Cristache, Senior Lecturer, DMD, PhD, Oral and Maxillofacial Surgeon, Project responsable, Carol Davila University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCDI-UEFISCDI 39/2018
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Chronic Periodontitis
Keywords: Melatonin; Hyaluronic Acid; Tetracycline; Metronidazole; topic paste; chronic periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetracycline-Metronidazole (TM) group (Active Comparator): Topical administration (in the periodontal pocket of affected teeth), for 30 consecutive days of 3%Tetracycline and 3%Metronidazole paste (TM), n=25 patients, considered control group.
  Interventions: Drug: Tetracycline-Metronidazole (TM) group
- TM-Melatonin-Hyaluronic acid (TM-MHa) group (Experimental): Topical administration (in the periodontal pocket of affected teeth), for 30 consecutive days of 3% Tetracycline, 3% Metronidazole, 0.18% Melatonin and 3% Hyaluronic Acid (TM-MHa) paste, n=25 patients, considered experimental group.
  Interventions: Drug: TM-Melatonin-Hyaluronic acid (TM-MHa) group

INTERVENTIONS:
Drug: Tetracycline-Metronidazole (TM) group — Following mechanical debridement (scaling and root planning) the above-mentioned paste will be topically administrated in the periodontal pocket of affected teeth once a day, for 30 consecutive days.
  Other Names: TM group
  Arms: Tetracycline-Metronidazole (TM) group
Drug: TM-Melatonin-Hyaluronic acid (TM-MHa) group — Following mechanical debridement (scaling and root planning) the above-mentioned paste will be topically administrated in the periodontal pocket of affected teeth once a day, for 30 consecutive days.
  Other Names: TM-MHa group
  Arms: TM-Melatonin-Hyaluronic acid (TM-MHa) group

SUMMARY:
The aim of the present study is to determine whether the association of Melatonin and Hyaluronic Acid to the antimicrobial TM paste (3% Tetracyclin and 3% Metronidazole) for periodontal maintenance therapy can improve the attachment level (AL) and alveolar bone support for moderate chronic periodontitis.

DETAILED DESCRIPTION:
Local drug delivery agents in periodontology has gained acceptance and popularity compared to systemic drugs due to decreased risk in development of resistant flora, opportunist infection, and side effects.

In order to improve the topical treatment for chronic periodontitis, Melatonin and Hyaluronic Acid have been added to antimicrobial topic paste commercially available.

* A complex matrix composed of Tetracycline, Metronidazole, Melatonin and Hyaluronic Acid have been developed for local treatment of chronic periodontitis.
* Microbiological, physical, chemical characterization of the newly obtained matrix and biocompatibility tests have been performed.
* A randomized clinical trial will be perform on 50 patients with moderate chronic periodontitis recruited based on eligibility criteria and informed consent signed.
* Mechanical debridement of the pockets by scaling and root planning will be performed prior to the adjunctive therapy.
* Extensive clinical examination including charting the remaining teeth, clinical attachment level (CAL), presence of dental plaque (PI), gingival index (GI), calculus (CI), bleeding on probing (BOP), radiographic assessment and identification of periodontal pathogens with micro-IDent® test will be performed at the beginning of the study and 6 month after its completion.
* Each patient will be randomized using sealed envelopes (according to a computer-generated randomization list) to one of the following topical administration (in the periodontal pocket of affected teeth), for 30 consecutive days: Tetracycline and Metronidazole paste (TM), n=25 patients and Tetracycline, Metronidazole, Melatonin, Hyaluronic Acid paste (TM-MHa), n=25 patients.
* A statistical evaluation of data recorded during the entire follow-up period will be performed.

ELIGIBILITY:
Inclusion Criteria:

* moderate chronic periodontitis, that is, > 2 interproximal sites with AL > 4 mm (not on the same tooth), or > 2 interproximal sites with pocket depth (PD) > 5 mm (not on the same tooth) (1),
* at least 20 teeth present in the mouth,
* no periodontal therapy during the last 6 months,
* no antibiotic during the last 6 months,
* good general health (no systemic condition affecting the course of periodontal disease, including malignancy), pregnancy,
* no allergy to the product components,
* good mental health.

Exclusion Criteria:

* Patients not willing to sign consent form.
* Patients not agreeing with the treatment protocol.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in Clinical attachment level (CAL) | before treatment (Baseline), at 6 months post treatment completion
  Changes CAL from Baseline (before treatment) at 6 months will be assessed using a standardised protocol.

SECONDARY OUTCOMES:
Changes in Alveolar bone height | before treatment (Baseline), at 6 months post treatment completion
  Changes in the alveolar bone height from Baseline (before treatment) at 6 months will be assessed using standardised Radiographic measurements.
Treatment's influence on bactrial pathogens | before treatment (Baseline), at 6 months post treatment completion
  Periodontal pathogens will be identified by performing micro-IDent® assay before treatment (Baseline) and 6 month after its completion. Micro-IDent® test uses chain polymerisation reaction, with colorimetric detection, to identify the following pathogens: Actinobacillus actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, Bacteroides forsythus, Treponema denticola.

CONTACTS AND LOCATIONS:
Overall Officials: CORINA MARILENA CRISTACHE, Principal Investigator — Carol Davila University of Medicine and Pharmacy
Locations (2):
- Romania (2):
  - Concordia Dent Clinic, Bucharest
  - "Carol Davila"University of Medicine and Pharmacy, Bucharest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eke PI, Page RC, Wei L, Thornton-Evans G, Genco RJ. Update of the case definitions for population-based surveillance of periodontitis. J Periodontol. 2012 Dec;83(12):1449-54. doi: 10.1902/jop.2012.110664. Epub 2012 Mar 16. PMID 22420873
- [Background] Feres M, Figueiredo LC, Soares GM, Faveri M. Systemic antibiotics in the treatment of periodontitis. Periodontol 2000. 2015 Feb;67(1):131-86. doi: 10.1111/prd.12075. PMID 25494600
- [Background] Matesanz-Perez P, Garcia-Gargallo M, Figuero E, Bascones-Martinez A, Sanz M, Herrera D. A systematic review on the effects of local antimicrobials as adjuncts to subgingival debridement, compared with subgingival debridement alone, in the treatment of chronic periodontitis. J Clin Periodontol. 2013 Mar;40(3):227-41. doi: 10.1111/jcpe.12026. Epub 2013 Jan 16. PMID 23320860
- [Background] Jepsen K, Jepsen S. Antibiotics/antimicrobials: systemic and local administration in the therapy of mild to moderately advanced periodontitis. Periodontol 2000. 2016 Jun;71(1):82-112. doi: 10.1111/prd.12121. PMID 27045432
- [Background] Koyama H, Nakade O, Takada Y, Kaku T, Lau KH. Melatonin at pharmacologic doses increases bone mass by suppressing resorption through down-regulation of the RANKL-mediated osteoclast formation and activation. J Bone Miner Res. 2002 Jul;17(7):1219-29. doi: 10.1359/jbmr.2002.17.7.1219. PMID 12096835
- [Background] Montero J, Lopez-Valverde N, Ferrera MJ, Lopez-Valverde A. Changes in crevicular cytokines after application of melatonin in patients with periodontal disease. J Clin Exp Dent. 2017 Sep 1;9(9):e1081-e1087. doi: 10.4317/jced.53934. eCollection 2017 Sep. PMID 29075409
- [Background] Andersen LP, Gogenur I, Rosenberg J, Reiter RJ. The Safety of Melatonin in Humans. Clin Drug Investig. 2016 Mar;36(3):169-75. doi: 10.1007/s40261-015-0368-5. PMID 26692007
- [Background] Diker N, Gulsever S, Koroglu T, Yilmaz Akcay E, Oguz Y. Effects of Hyaluronic Acid and Hydroxyapatite/Beta-tricalcium Phosphate in Combination on Bone Regeneration of a Critical-size Defect in an Experimental Model. J Craniofac Surg. 2018 Jun;29(4):1087-1093. doi: 10.1097/SCS.0000000000004338. PMID 29438204
- [Background] Pirnazar P, Wolinsky L, Nachnani S, Haake S, Pilloni A, Bernard GW. Bacteriostatic effects of hyaluronic acid. J Periodontol. 1999 Apr;70(4):370-4. doi: 10.1902/jop.1999.70.4.370. PMID 10328647
- [Background] Sakai A, Akifusa S, Itano N, Kimata K, Kawamura T, Koseki T, Takehara T, Nishihara T. Potential role of high molecular weight hyaluronan in the anti-Candida activity of human oral epithelial cells. Med Mycol. 2007 Feb;45(1):73-9. doi: 10.1080/13693780601039607. PMID 17325947